CLINICAL TRIAL: NCT04546204
Title: COMPARISON OF OBSTETRIC AND NEONATAL OUTCOMES BETWEEN SYRIAN ADOLESCENT REFUGEES AND LOCAL TURKISH ADOLESCENT CITIZENS.
Brief Title: COMPARISON OF OBSTETRIC AND NEONATAL OUTCOMES OF ADOLESCENT PREGNANCİES
Status: Completed | Type: Observational
Sponsor: Alkü Alanya Education and Research Hospital (Other)
Responsible Party: Principal Investigator, MERAL TUĞBA ÇİMŞİR, Assistant Professor, Alkü Alanya Education and Research Hospital
Other Study IDs: adolescentpregnancy
Record Dates: First submitted 2020-09-06; First posted 2020-09-11 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Adolescent Development; Pregnancy Related

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: vaginal delivery — normal vaginal spontaneous delivery

SUMMARY:
ABSTRACT

Adolescent pregnancy rates are gradually increasing in the recent decades. As a reason of war nutritional difficulties, language differences and difficulty in applying to the health institution causes lack of prenatal care. As a reason of absence of prenatal care, associated medical complications can occur. 525 adolescent women who gave birth to singletons agreed to participate in this study. Data on maternal demographic and obstetric characteristics as well as neonatal outcomes were analyzed. In conclusion, adolescent pregnancy continues to be an important social problem due to the health support needs. However, the results of our present study are important in terms of showing that the perinatal care is quietly improved in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* 14-16 y Age

Exclusion Criteria:

* over 16 years

Ages: 14 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: adolescent pregnancy outcomes
Sampling Method: Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
vaginal delivery rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Alkü Education and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No